CLINICAL TRIAL: NCT00797771
Title: Evaluation of User Satisfaction Using the ADI Insulin Pump
Brief Title: User Satisfaction Using the ADI Insulin Pump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NiliMedix (Industry)
Responsible Party: Dr. Hanna Levy, NiliMedix
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NM-HU-01
Record Dates: First submitted 2008-11-23; First posted 2008-11-25 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes
Keywords: Insulin delivery
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): "Adi" insulin pump users
  Interventions: Device: "Adi" Insulin pump

INTERVENTIONS:
Device: "Adi" Insulin pump — insulin delivery will be defined by the physician

SUMMARY:
Approximately 250,000 people worldwide are currently being treated with an insulin pump. This number is growing dramatically as these devices become smaller and more user-friendly. Insulin pumps allow for tight metabolic control and lifestyle flexibility while minimizing the number of hypoglycemic events.

The NiliMedix ADI Insulin Pump is an ambulatory, battery operated, rate programmable micro- infusion pump, designed for continuous delivery of insulin. A custom reservoir is driven by the pressure of insulin within it to deliver preset basal profiles and patient programmed bolus of insulin through custom infusion sets, into subcutaneous tissue.

This type of device requires extensive user interaction and education in order to ensure its safety. This study was designed to test the independent home-use of the NiliMedix ADI Insulin Pump, and to evaluate user's satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Male/female age 18 years and up.
* Subject is diagnosed as Type 1 Diabetes.
* Pump Users for at least 6 months
* HbA1c: less than 8.5%
* Capable of reading pump screens in English.
* Subject understands the study procedure.
* Subject is willing to sign the informed consent form and comply with the study requirements.

Exclusion Criteria:

* Major physical, motor, mental, behavioral, or psychiatric limitations.
* Subject experienced a severe hypoglycemic episode that led to hospitalization during the last 6 months.
* Subject experienced an episode of Ketoacidosis during the last 6 months, while using an insulin pump.
* Concurrent additional major illness.
* Subject objects to the study protocol.
* Physician objection
* Concurrent participation in other study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
User satisfaction regarding the "Adi" pump functioning will be evaluated by questionnaire. The questionnaire will be administrated during the last study visit | End of study

SECONDARY OUTCOMES:
Number of severe hypoglycemic events | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Shalitin, MD, Principal Investigator — Schnieder Children's Medical Center Israel
Locations (1):
- Schnieder Children's Medical Center, Petah Tikva, Israel